CLINICAL TRIAL: NCT04408235
Title: Randomised Controlled Trial Comparing High Versus Low LMWH Dosages in Hospitalized Patients With Severe COVID-19 Pneumonia and Coagulopathy Not Requiring Invasive Mechanical Ventilation
Brief Title: High Versus Low LMWH Dosages in Hospitalized Patients With Severe COVID-19 Pneumonia and Coagulopathy
Acronym: COVID-19 HD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Marco Marietta, Head, Hemostasis and Thrombosis Unit, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT N°: 2020-001972-13
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: COVID; Pneumonia, Viral; Coagulation Disorder
Keywords: COVID-19; PNEUMONIA; COAGULOPATHY; LOW-MOLECULAR WEIGHT HEPARIN; ENOXAPARIN
MeSH Terms: conditions — Pneumonia, Viral; Hemostatic Disorders; COVID-19; Pneumonia | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: This is a multicentre, randomised controlled, open label, investigator sponsored, two arms study.
Who Masked: Investigator
Masking Description: Randomisation will be centrally performed by using a secure, web-based system, which will be developed by the Methodological and Statistical Unit at the Azienda Ospedaliero-Universitaria of Modena. Randomisation stratified by 4 factors: 1) Gender (M/F); 2) Age (<75/≥75 years); 3) BMI (<30/≥30); 4) Co-morbidities (0-1/>2) with random variable block sizes will be generated by STATA software. The web-based system will guarantee the allocation concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Dose LMWH (Active Comparator): Enoxaparin 4000 IU daily
  Interventions: Drug: Enoxaparin
- High-Dose LMWH (Experimental): Enoxaparin 70 IU/kg twice daily
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Low-Dose LMWH: enoxaparin 4000 IU daily; High dose LMWH: 70 IU/kg twice daily
  Other Names: Inhixa®

SUMMARY:
Randomized, controlled study conducted in hospitalized patients with severe COViD-19 pneumonia and coagulopathy not requiring invasive mechanical ventilation.

Aim of this study is to assess whether high doses of Low Molecular Weight Heparin (LMWH) (ie. Enoxaparin 70 IU/kg twice daily) compared to standard prophylactic dose (ie, Enoxaparin 4000 IU once day) are:

1. More effective to prevent clinical worsening, defined as the occurrence of at least one of the following events, whichever comes first, during hospital stay:

   1. Death
   2. Acute Myocardial Infarction [AMI]
   3. Objectively confirmed, symptomatic arterial or venous thromboembolism [TE]
   4. Need for either non-invasive - Continuous Positive Airway Pressure (Cpap) or Non-Invasive Ventilation (NIV) - or invasive mechanical ventilation for patients who are in standard oxygen therapy by delivery interfaces at randomisation
   5. Need for invasive mechanical ventilation for patients who are in non-invasive mechanical ventilation at randomisation
2. Similar in terms of major bleeding risk during hospital stay

DETAILED DESCRIPTION:
This is a multicentre, randomised controlled, open label, investigator sponsored, two arms study.

The study will involve 7 Italian Academic and non-Academic Internal Medicine Units, 2 Infectious Diseases Units, 1 Respiratory Diseases Unit.

Patients who satisfy all inclusion criteria and do not have any exclusion criteria and have signed written informed consent, will be randomly assigned to a Low-Dose LMWH group (Control Group) or High-Dose LMWH group (Intervention Group) in a 1:1 ratio.

Control Group (Low-Dose LMWH): patients in this group will be administered Enoxaparin (Inhixa®) at standard prophylactic dose (i.e., 4000 IU subcutaneously once day).

Intervention Group (High-Dose LMWH): patients in this group will be administered Enoxaparin (Inhixa®) at dose of 70 IU/kg every 12 hours, as reported in the following table.

The study is conceived as open-label: patients and all health-care personnel involved in the study will be aware of the assigned group.

The treatments will be initiated as soon as possible after randomization (maximum allowed starting time 12h after randomization).

Patients allocated to the two arms will maintain the doses of Enoxaparin, as stated in the protocol, until:

1. hospital discharge or
2. when at least one of the following events occurs:

   1. Acute Myocardial Infarction [AMI]
   2. Objectively confirmed, symptomatic arterial or venous thromboembolism [TE]
   3. Need for either non-invasive - Continuous Positive Airway Pressure (Cpap) or Non-Invasive Ventilation (NIV) - or invasive mechanical ventilation for patients, who are in standard oxygen therapy by delivery interfaces at randomisation
   4. Need for invasive mechanical ventilation for patients, who are in non-invasive mechanical ventilation at randomisation
   5. Major bleeding
   6. Any adverse events and clinical condition requiring interruption of the scheduled intervention according to the judgement of the physician in charge
   7. Death

The decision about what type and dose of antithrombotic treatment to administer, after the interruption of assigned dose of Enoxaparin, will be left to clinical judgement of the physicians in charge.

Any information about the type and dose of antithrombotic treatments administered after the interruption of the assigned dose of Enoxaparin will be collected until the hospital discharge or death.

Each patient will be followed-up until hospital discharge. Information about the status (dead/alive) of patients who are discharged from hospital before 30 days will be sought on Day 30 from randomisation.

ELIGIBILITY:
Inclusion Criteria (all required):

* Positive SARS-CoV-2 diagnostic (on pharyngeal swab of deep airways material)
* Severe pneumonia defined by the presence of at least one of the following criteria:

  1. Respiratory Rate ≥25 breaths /min
  2. Arterial oxygen saturation≤93% at rest on ambient air
  3. PaO2/FiO2 ≤300 mmHg
* Coagulopathy, defined by the presence of at least one of the following criteria:

  1. D-dimer >4 times the upper level of normal reference range
  2. Sepsis-Induced Coagulopathy (SIC) score >4
* No need for invasive mechanical ventilation

Exclusion Criteria:

* Invasive mechanical ventilation
* Thrombocytopenia (platelet count < 80.000 mm3)
* Coagulopathy: INR >1.5, aPTT ratio > 1.4
* Impaired renal function (eGFR calculated by CKD-EPI Creatinine equation < 30 ml/min)
* Known hypersensitivity to enoxaparin
* History of heparin induced thrombocytopenia
* Presence of an active bleeding or a pathology susceptible of bleeding in presence of anticoagulation (e.g. recent haemorrhagic stroke, peptic ulcer, malignant cancer at high risk of haemorrhage, recent neurosurgery or ophthalmic surgery, vascular aneurysms, arteriovenous malformations)
* Concomitant anticoagulant treatment for other indications (e.g. atrial fibrillation, venous thromboembolism, prosthetic heart valves).
* Concomitant double antiplatelet therapy
* Administration of therapeutic doses of LMWH, fondaparinux, or unfractionated heparin (UFH) for more than 72 hours before randomization; prophylactic doses are allowed
* Pregnancy or breastfeeding or positive pregnancy test
* Presence of other severe diseases impairing life expectancy (e.g. patients are not expected to survive 28 days given their pre-existing medical condition)
* Lack or withdrawal of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Clinical worsening, defined as the occurrence of at least one of the following events, whichever comes first: | through study completion, up to 30 days
  1. Death
  2. Acute Myocardial Infarction [AMI]
  3. Objectively confirmed, symptomatic arterial or venous thromboembolism [TE]
  4. Need for either non-invasive - Continuous Positive Airway Pressure (Cpap) or Non-Invasive Ventilation (NIV) - or invasive mechanical ventilation for patients, who are in standard oxygen therapy by delivery interfaces at randomisation
  5. Need for invasive mechanical ventilation for patients, who are in non-invasive mechanical ventilation at randomisation

SECONDARY OUTCOMES:
Any of the following events occurring within the hospital stay | through study completion, up to 30 days
  1. Death
  2. Acute Myocardial Infarction [AMI]
  3. Objectively confirmed, symptomatic arterial or venous thromboembolism [TE]
  4. Need for either non-invasive - Continuous Positive Airway Pressure (Cpap) or Non-Invasive Ventilation (NIV) - or invasive mechanical ventilation for patients, who are in standard oxygen therapy by delivery interfaces at randomisation
  5. Need for invasive mechanical ventilation for patients, who are in non-invasive mechanical ventilation at randomisation
  6. Improvement of laboratory parameters of disease severity, including:
     * D-dimer level
     * Plasma fibrinogen levels
     * Mean Platelet Volume
     * Lymphocyte/Neutrophil ratio
     * IL-6 plasma levels
Mortality at 30 days | 30 days
  Information about patients' status will be sought in those who are discharged before 30 days on Day 30 from randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Marietta, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena
Locations (1):
- Azienda Ospedaliero-Universitaria, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Leisman DE, Deutschman CS, Legrand M. Facing COVID-19 in the ICU: vascular dysfunction, thrombosis, and dysregulated inflammation. Intensive Care Med. 2020 Jun;46(6):1105-1108. doi: 10.1007/s00134-020-06059-6. Epub 2020 Apr 28. No abstract available. PMID 32347323
- [Background] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Marietta M, Ageno W, Artoni A, De Candia E, Gresele P, Marchetti M, Marcucci R, Tripodi A. COVID-19 and haemostasis: a position paper from Italian Society on Thrombosis and Haemostasis (SISET). Blood Transfus. 2020 May;18(3):167-169. doi: 10.2450/2020.0083-20. Epub 2020 Apr 8. No abstract available. PMID 32281926
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Background] Thachil J. The versatile heparin in COVID-19. J Thromb Haemost. 2020 May;18(5):1020-1022. doi: 10.1111/jth.14821. Epub 2020 Apr 27. No abstract available. PMID 32239799
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773